CLINICAL TRIAL: NCT02023593
Title: Phase Ⅱ Study of FOLFIRI as Second-Line Chemotherapy for Metastatic Esophageal Carcinoma
Brief Title: FOLFIRI as Second Line Chemotherapy for Metastatic Esophageal Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yuhong Li (Other)
Responsible Party: Sponsor-Investigator, Yuhong Li, MD,Ph D, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FOLFIRI-29
Record Dates: First submitted 2013-12-16; First posted 2013-12-30 (Estimated); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Advanced Esophageal Carcinoma
MeSH Terms: interventions — IFL protocol; Irinotecan; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FOLFIRI (Experimental): Patients will receive FOLFIRI every 2 weeks: Irinotecan 180mg/m2 IV over 90 minutes on Day 1; Leucovorin IV over 2 hours on Day 1(l-LV 200 mg/m2 or dl-LV 400 mg/m2 ); 5-Fluorouracil 400 mg/m2 IV bolus on Day 1; followed by 5-Fluorouracil 2.4 g/m2 for 46 hours continuous infusion.
  Interventions: Drug: FOLFIRI

INTERVENTIONS:
Drug: FOLFIRI — Patients will receive FOLFIRI every 2 weeks: Irinotecan 180mg/m2 IV over 90 minutes on Day 1; Leucovorin IV over 2 hours on Day 1(l-LV 200 mg/m2 or dl-LV 400 mg/m2 ); 5-Fluorouracil 400 mg/m2 IV bolus on Day 1; followed by 5-Fluorouracil 2.4 g/m2 for 46 hours continuous infusion.
  Other Names: Irinotecan; Leucovorin; 5-Fluorouracil

SUMMARY:
This phase Ⅱ study was designed to evaluate the efficacy and safety of FOLFIRI as second-line treatment for metastatic esophageal carcinoma.

DETAILED DESCRIPTION:
Although there are no standard second-line treatment for metastatic esophageal carcinoma, some studies have showed that irinotecan, fluorouracil may be effective in treating patients with metastatic esophageal carcinoma after failure of first-line treatment. Since irinotecan, fluorouracil, and leucovorin work in different ways to stop the growth of tumor. Giving more than one drug may be more effective. In this phase Ⅱ trial, the investigator would like to observe the efficacy and safety of FOLFIRI(Irinotecan/5-FU/leucovorin ) as second-line treatment for metastatic esophageal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients have provided a signed Informed Consent Form
* Karnofsky score ≥70
* Age: 18-75 years old
* Histologically confirmed diagnosis of advanced esophageal carcinoma
* Patients have Received and progressed on first-line treatment, and not received CPT-11 or Fluoropyrimidine based palliative chemotherapy
* Measurable disease in at least 1 diameter by CT scan or MRI as per RECIST 1.1 criteria
* Life expectancy ≥ 3 months
* Patient has adequate bone marrow and organ function

  * Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/L
  * Platelets ≥ 75 x 109/L
  * Hemoglobin ≥ 9.0 g/dL
* Patient has adequate liver function

  * AST and ALT not more than 2.5 times ULN (not more than 5.0 times ULN if there is liver metastasis)
  * Serum bilirubin ≤ 2 x ULN
* Creatinine ≤ 1.5 times ULN
* Good compliance

Exclusion Criteria:

* Pregnant or lactating women
* Brain metastasis or only with bone metastasis.
* Patients with severe infection or active peptic ulcer which need treatment
* Severe systemic disease out of control such as unstable or uncompensated respiratory, cardiac, liver, renal diseases
* Patient has a concurrent malignancy or has a malignancy within 5 years of study enrollment, (with the exception of non-melanoma skin cancer or cervical carcinoma in situ
* Psychiatric illness that would prevent the patient from giving informed consent
* Patient is concurrently using other approved or investigational antineoplastic agent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Disease control rate | Up to 24 weeks

SECONDARY OUTCOMES:
Overall survival | From the date of first drug administration until the date of death, assessed up to 60months
Adverse events | Each follow up visit, assessed up to 24 weeks
  Safety profile will be assessed using the NCI CTCAE version 3.0
Progression free survival | From the date of first drug administration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Li Yuhong, Ph D, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China